CLINICAL TRIAL: NCT03824184
Title: Endometrial Assessment Women With Infertility Who Will do IUI and ICSI
Brief Title: Endometrial Assessment of Women With Uterine Infection
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Aljazeera Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Uterine infection
Record Dates: First submitted 2019-01-28; First posted 2019-01-31 (Actual); Last update posted 2023-09-26 (Actual); Status verified 2023-09

CONDITIONS: Infertility
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Intervention Model Description: A randomized controlled trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hysteroscopic evaluation (Active Comparator): Hysteroscopic evaluation Active group : infection Manipulation of endometrium with saline
  Interventions: Procedure: manipulation of endometrium
- control group (Other): Hysteroscopic evaluation Control group : No infection
  Interventions: Procedure: manipulation of endometrium

INTERVENTIONS:
Procedure: manipulation of endometrium — Manipulation of endometrium with saline
  Other Names: Saline infusion

SUMMARY:
Unexplained infertility is clinically diagnosed when there are no apparent or clear factors causing infertility on regular infertility assessment tools . Failure of implantation is a possible factor causing unexplained infertility .

DETAILED DESCRIPTION:
Implantation is the main rate limiting step in IVF outcome. Implantation is described at the cellular and the molecular levels by adhesion or fixation of a good quality embryo to receptive endometrium within a critical period of time, which is called the window of implantation

ELIGIBILITY:
Inclusion Criteria:

* Women with infertility age from 20-40 years

Exclusion Criteria:

* Any factor of infertility

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — infertile women
Enrollment: 300 (Estimated)
Dates: Start 2019-02-02 (Actual); Primary Completion 2024-05-03 (Estimated); Study Completion 2024-06-20 (Estimated)

PRIMARY OUTCOMES:
the number of women who will get pregnant after IUI | within 4 weeks
  How many women will get pregnant after IUI

CONTACTS AND LOCATIONS:
Overall Officials: Mahmoud Alalfy, Principal Investigator — Algazeerah hospital -Location (Giza -Egypt ) and National Research centre egypt
Locations (1):
- Algazeerah and Kasralainy hospital, Giza, Egypt

IPD SHARING:
Plan to Share IPD: No